CLINICAL TRIAL: NCT03747146
Title: Expanding the Peri-operative Surgical Home Model: ERAS TKR With a Transitional Pain Service (TeleTPS)- Continuous Adductor Canal Catheter Versus Adductor Canal Block for Total Knee Arthroplasty, a Randomized Double-blind Controlled Trial
Brief Title: Enhanced Recovery After Surgery (ERAS) Total Knee Replacement (TKR) With a Transitional Pain Service
Acronym: EKAT-TeleTPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-1858
Record Dates: First submitted 2018-11-06; First posted 2018-11-20 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Continuous Adductor Canal Catheter (ACC) (Active Comparator): Patients will receive a combined spinal epidural, PAI, IPACK, and a continuous adductor canal catheter
  Interventions: Device: Continuous Adductor Canal Catheter (ACC)
- Adductor Canal block with sham catheter (Sham Comparator): Patients will receive a combined spinal epidural, PAI, IPACK, and an adductor canal block. The patient will also receive a sham catheter.
  Interventions: Device: Adductor Canal block with sham catheter

INTERVENTIONS:
Device: Continuous Adductor Canal Catheter (ACC) — At the end of the case or in the PACU, a pseudo sham catheter will be affixed mid-thigh to the skin using dermabond, steri-strips, and a chg tegaderm dressing. The catheter will be connected to the disposable pump filled with sterile saline (400 cc) and the flow rate will be set to 0. The pump will be enclosed in a carrier bag provided by the company. To ensure blinding, the carrier bag will be taped to prevent the patient from accessing it.
  Arms: Continuous Adductor Canal Catheter (ACC)
Device: Adductor Canal block with sham catheter — Adductor canal block (ACB) will be administered. At the end of the case or in the PACU, a catheter will be inserted and affixed mid-thigh to the skin using dermabond, steri-strips, and a chg tegaderm dressing. The catheter will be connected to the disposable pump filled with sterile saline (400 cc) and the flow rate will be set to 0. The pump will be enclosed in a carrier bag provided by the company. To ensure blinding, the carrier bag will be taped to prevent the patient from accessing it.
  Arms: Adductor Canal block with sham catheter

SUMMARY:
A comparison of two anesthetic techniques for total knee replacements: (1) Peri-Articular Injection (PAI), local infiltration between the popliteal artery and capsule of the knee block (IPACK) and single-shot adductor canal block (ACB) vs. (2) PAI, IPACK and continuous adductor canal block catheter (ACC).

DETAILED DESCRIPTION:
Patients will be randomized to one of two groups: one group will receive a PAI, IPACK and single-shot adductor canal block; one group will receive PAI, IPACK and continuous adductor canal block catheter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with osteoarthritis scheduled for a primary total knee arthroplasty with a participating surgeon
* Planned use of regional anesthesia
* Ability to follow study protocol
* English speaking (secondary outcomes include questionnaires validated in English only)
* Lives within one hour of the hospital
* Has a smart phone

Exclusion Criteria:

* Hepatic or renal insufficiency
* Younger than 18 years old or older than 65 years ol
* Patients undergoing general anesthesia
* Allergy or intolerance to one of the study medications
* BMI >40
* Diabetes
* American Society of Anesthesiologists (ASA) status III or IV
* Chronic gabapentin/pregabalin use (regular use for longer than 3 months)
* Patients with chronic pain (from a referral to chronic pain service) or a pain catastrophizing scale (PCS >30)
* Patients with severe valgus deformity or flexion contracture
* Patients unable to follow home catheter instructions and unwilling to go home with an infusing catheter
* Patients who have no home caregivers in the event that a catheter is to be sent home with the patient
* Patients with planned stay at rehab facility (to avoid medical device being tampered with at the rehab facility)
* Non-English speakers (secondary outcomes include questionnaires validated in English only)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2018-11-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption during 24-48 hour period | Post-operative day 1-2 (24-48 hours post spinal induction)
  Patients will be asked to report their opioid consumption during the 24-48 hour time period after spinal induction. This data will be converted to morphine milligram equivalents (mme).

SECONDARY OUTCOMES:
Opioid consumption during post-anesthesia care unit (PACU) stay | Day of surgery from PACU arrival until transfer to in-patient floor (up to 48 hours)
  Patients will be asked to report their opioid consumption during their stay in the post-anesthesia care unit. This data will be converted to morphine milligram equivalents (mme).

CONTACTS AND LOCATIONS:
Overall Officials: David Kim, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No